CLINICAL TRIAL: NCT01912144
Title: Bioavailability of Coffee Phenolic Acids and Cardiovascular Health in Healthy Humans.
Brief Title: Absorption of Phenolic Acids From Coffee in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Gary Williamson, Prof, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MEEC 10-035
Record Dates: First submitted 2013-07-17; First posted 2013-07-30 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Bioavailability; Cardiovascular Health Status
MeSH Terms: interventions — Coffee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- coffee (Other): Coffee beverage
  Interventions: Other: Coffee

INTERVENTIONS:
Other: Coffee

SUMMARY:
Phenolic acids are naturally-occurring constituents of plant-derived foods and beverages and are characterised by a phenol ring in their structure. The phenolic compounds we are going to focus on in this study are the Chlorogenic acids (CGAs), a family of esters conjugates formed between a Hydroxycinnamic acid and quinic acid (1) and that show a strong antioxidant activity (2).

HCAs represent about 50% of the total polyphenolic coumpounds intake in a typical UK diet (3) and for people who drink it, coffee is a/the major dietary source of/for HCAs (4). A few studies suggest protective effects for cardiovascular diseases (5), neurodegenerative diseases, type 2 diabetis and liver and kidneys cancer risk. However, many data in the field are obtained from in vitro and/or in animal, and it is difficult and dangerous to extrapolate between these and risk in humans of development or progression of particular health conditions, more human studies are therefore needed.

We aim to compare people that metabolise the best CGAs from coffee to those that metabolise them the least well. This will be achieved by measuring the metabolites in urine. The effect of CGAs on the human body does not only depend on the amount ingested, but also on the quality of the metabolism, we therefore also want to determine which mechanisms are responsible for inter-individual variations in order to identify any link with health biomarkers, these including non-cellular inflammation and cardiovascular risk indicators.

For this cohort study funded by the University of Leeds, approximately 60 healthy volunteers will be recruited at the School of Food Science & Nutrition. If they meet the selection criteria, participants will be asked to undergo a 36-hour wash-out period. During those 36 hours, participants won't be allowed to drink coffee, they will be asked to follow a diet low in phenolic acids and keep a record of their meals. On the first day of the study, a single dose of coffee rich in antioxidants will be given to the participant and urine will be collected from that time until 36 hours after coffee consumption. Participants will be followed again after 5 to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Normal Body Mass Index (BMI) 18-29 kg/m2
* Non-smoker, former or weak smoker (max. 5 cigarettes per day)
* No more than 4 alcoholic units as a regular and daily consumption

Exclusion Criteria:

* diagnosed chronic disease (e.g. pancreas, kidneys, liver, heart)
* haemophilia
* long term prescribed medication (contraceptive medication allowed)
* previous GI (gastrointestinal) tract operation
* pregnant or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Quantitative absorption of chlorogenic acids metabolites | up to 7 months
  Analysis using liquid chromatography with or without mass spectrometry, colorimetric and enzyme-linked immunosorbent assays.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Williamson, PhD, Principal Investigator — University of Leeds
Locations (1):
- School of Food Science, University of Leeds, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Background] M.N. Clifford, J. Sci. Food Agric. 80 (2000) 1033-1043.] [Clifford MN, Chlorogenic acids and other cinnamates-nature, occurrence and dietary burden. Journal of the Science of Food and Agriculture 1999, 79(3), 362-372
- [Background] Stalmach et al. 2006, On-line HPLC analysis of the antioxidant activity of phenolic compounds in brewed paper-filtered coffee. Brasil J Plant Physiol 18:253-262
- [Background] Stevenson DE, Hurst RD. Polyphenolic phytochemicals--just antioxidants or much more? Cell Mol Life Sci. 2007 Nov;64(22):2900-16. doi: 10.1007/s00018-007-7237-1. PMID 17726576
- [Background] D'Archivio M, Filesi C, Di Benedetto R, Gargiulo R, Giovannini C, Masella R. Polyphenols, dietary sources and bioavailability. Ann Ist Super Sanita. 2007;43(4):348-61. PMID 18209268
- [Background] Stanner 2005, Cardiovascular disease: Diet, Nutrition and emerging risk factors. The report of the british nutrition foundation task force. Blackwell Science for the British nutrition foundation: Oxford, UK